CLINICAL TRIAL: NCT02797899
Title: Effect of Platelet Rich Fibrin Palatal Bandage on Pain Scores and Wound Healing After Free Gingival Graft
Brief Title: Effect of PRF Palatal Bandage on Pain Scores and Wound Healing After Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maha A. Bahammam, Associate Professor and Consultant of Periodontology, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 285/254/1434
Record Dates: First submitted 2016-06-02; First posted 2016-06-14 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Pain; Wound Healing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palatal donor site received PRF (Active Comparator): Following profound anesthesia and harvesting free gingival graft from the palate, the graft was positioned to the recipient area. The donor area were cleaned with sterile saline and received platelet rich fibrin and periodontal pack as assigned randomly by a flip of coin during the screening visits.
  Interventions: Device: Platelet Rich Fibrin
- Palatal donor site NOT receiving PRF (Active Comparator): Following profound anesthesia and harvesting free gingival graft from the palate, the graft was positioned to the recipient area. The donor area were cleaned with sterile saline and sutured followed by periodontal pack application.
  Interventions: Device: Platelet Rich Fibrin

INTERVENTIONS:
Device: Platelet Rich Fibrin — Native growth factors

SUMMARY:
Background: Free gingival graft (FGG) is used to increase keratinized tissue dimensions. This prospective clinical trial was conducted aiming to determine whether the addition of an autologous platelet-rich fibrin (PRF) would improve soft tissue healing of donor sites and decrease pain scores.

Methods: Twenty four patients were planned to receive FGG to augment keratinized tissue dimensions in the mandibular incisors area. Donor sites were assigned randomly to receive PRF or not by a flip of a coin during the screening visit. Patients were instructed to complete a pain study form. The palatal donor area were evaluated for complete wound healing records. These data were assessed and recorded before surgery, and 1,2,3,4 and 8 weeks postoperatively.

DETAILED DESCRIPTION:
Background: Despite a relatively painful surgical procedure, free gingival graft (FGG) is still commonly used to increase keratinized tissue dimensions. This prospective clinical trial was conducted aiming to determine whether the addition of an autologous platelet-rich fibrin (PRF) after harvesting a FGG would improve soft tissue healing of donor sites and subsequently decrease pain scores.

Methods: Twenty four patients were planned to receive FGG to augment keratinized tissue dimensions in the mandibular incisors area. Enrolled patients received periodontal examination, oral hygiene instructions and full-mouth debridement followed by standardized FGG of similar dimensions. Donor sites were assigned randomly to receive PRF or not by a flip of a coin during the screening visit. Patients were instructed to complete a pain study form to analyze pain scores including VAS, NRS-101, VRS-4 as well as three anxiety scales at base line. The palatal donor area were evaluated for complete wound healing based on the degree of color match, tissue texture, and contour of the surgical area compared to preoperative records. These data were assessed and recorded before surgery, and 1,2,3,4 and 8 weeks postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* lack of keratinized tissue in the mandibular central incisor region

Exclusion Criteria:

* smoking
* uncontrolled systemic disease that might contraindicate periodontal surgery
* severe gag reflex preventing maxillary surgical procedure
* inability or unwillingness to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes in Visual Analog scale (VAS) | 1, 2, 3, 4 and 8 weeks
  a visual analog scale (VAS) consisting a 10-cm line with two extremes at either end. "no pain" and "pain that could not be more severe". Patients were asked to mark a point on the line that represent their level of perceived pain

SECONDARY OUTCOMES:
Changes in contour of the surgical area | 1, 2, 3, 4 and 8 weeks
  To check for wound healing; contour of the surgical area was examined and compared to preoperative records
Changes in degree of color match | 1, 2, 3, 4 and 8 weeks
  To check for wound healing; degree of color match was examined and compared to preoperative records
Changes in tissue texture | 1, 2, 3, 4 and 8 weeks
  To check for wound healing; tissue texture was examined and compared to preoperative records

IPD SHARING:
Plan to Share IPD: No